CLINICAL TRIAL: NCT04973527
Title: A Phase I, Multicenter Study to Evaluate the Safety, Tolerability, and Efficacy of LCAR-T2C CAR-T Cells in Relapsed or Refractory CD4+ T Lymphocyte Tumor Patients
Brief Title: LCAR-T2C CAR-T Cells in Relapsed or Refractory CD4+ T Lymphocyte Tumor
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Both the sponsors and collaborator are considering terminating the study
Sponsor: Beijing Boren Hospital (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRYY-IIT-LCYJ-2021-011
Record Dates: First submitted 2021-07-07; First posted 2021-07-22 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: T Cell Lymphoma; T-cell Leukemia
MeSH Terms: conditions — Lymphoma, T-Cell; Leukemia, T-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCAR-T2C CAR-T cells in relapsed or refractory CD4+ T lymphocyte tumor (Experimental): An open label, multi center, single arm Phase I study to evaluate the safety, tolerability, and efficacy of LCAR-T2C CAR-T cells in relapsed or refractory CD4+ T lymphocyte tumor.
  Interventions: Drug: Efficacy of LCAR-T2C CAR-T cells

INTERVENTIONS:
Drug: Efficacy of LCAR-T2C CAR-T cells — CD4-directed CAR-T cells administered with lymphoid depletion, and to obtain the preliminary efficacy results in subjects who have been diagnosed with relapsed or refractory CD4 positive T lymphocyte tumor

SUMMARY:
This is a multicenter phase I clinical study evaluating the safety, tolerability, and efficacy of LCAR-T2C cell agents targeting CD4 in patients with relapsed/refractory CD4-positive T lymphocytic tumors. Thirty-three subjects will be enrolled. Subjects will be pretreated with chemotherapy prior to infusion of CAR T cells: about 5 days before cells transfusion, the patients who planned to reinfuse CAR T cells were treated with fluorodarabine 30 mg/m2( body surface area) and cyclophosphamide 300 mg/m2( body surface area) for 3 days. hen this study will be using a 3+3 dose escalation approach from dose 1 (DL-1): 5×105 to dose 2 (dl-2): 1.5×106 , to dose 3 (dl-3): 5×106 to dose 4 (dl-4): 10.0×106. Below the lowest dose was reinfused at the PI's discretion.

DETAILED DESCRIPTION:
This is an open, dose escalation/dose extension study of LCAR-T2C CAR-T cells administered to patients with T lymphocyte tumor. The aim of the study is to evaluate the safety, tolerability, and efficacy of LCAR-T2C CAR-T cells. The auto-CAR-T cells will be infused in single-dose.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF)
2. Age 18 Years to 75 Years
3. Pathological diagnosis of refractory/relapsed CD4+ T lymphocyte tumor (one of the following):

   a. T-cell Non-Hodgkin lymphoma(T-NHL)：The best response is progressive disease(PD) or stable disease(SD) after at least 1 prior line of therapy（at least 2 complete cycle of therapy） b. T-cell Acute lymphoblastic leukemia(T-ALL)：The best response is not complete response(CR) after induction therapy
4. Measurable disease is necessary at Screening
5. Life expectancy ≥ 3 months
6. Eastern Cooperative Oncology Group (ECOG) Performance Status grade of 0 -2.

The screening phase clinical laboratory values meet the following criteria. Laboratory test(s) may be repeated once, to determine if the subject qualifies for study participation :

Blood routine:

HGB≥6g/dL；PLT≥20×10^9/L; ANC≥1.0×10^9/L; LY≥0.3×10^9/L

Blood biochemical parameters:

1. Aspartate and alanine aminotransferases (AST, ALT) ≤ 2.5 times ULN (in the presence of liver metastasis, AST and ALT≤5 times ULN)
2. Serum creatinine (Scr) ≤ 1.5 times ULN, estimated glomerular filtration rate (eGFR) > 60mL/min (only when Scr>1.5 times ULN)
3. Total bilirubin ≤ 1.5 times of the normal upper limit (ULN)
4. International Normalized Ratio (INR) ≤ 1.5 times ULN, PT≤ 1.5 times ULN, APTT≤ 1.5 times ULN

Exclusion Criteria:

1. Prior treatment with CAR-T therapy directed at any target.
2. Any therapy that is targeted to CD4.
3. Prior treatment with an allogeneic stem cell transplant
4. Any malignancy besides the T lymphocyte tumor categories under study, exceptions include

   1. Any other malignancy curatively treated and disease-free for at least 2 years prior to enrollment
   2. History of non-melanoma skin cancer with sufficient treatment and currently no evidence of recurrence
5. Those who are positive for any index of hepatitis B surface antigen (HBsAg), hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C antibody (HCV-Ab), hepatitis C virus ribonucleic acid (HCV RNA), and human immunodeficiency virus antibody (HIV-Ab)
6. The following cardiac conditions:

   1. New York Heart Association (NYHA) stage III or IV congestive heart failure
   2. Myocardial infarction or coronary artery bypass graft (CABG) 6 months prior to enrollment
   3. History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
   4. History of severe non-ischemic cardiomyopathy
   5. Impaired cardiac function (LVEF <45%) as assessed by echocardiogram or multiple-gated acquisition (MUGA) scan (performed ≤8 weeks of apheresis)

Prior antitumor therapy as follows, prior to apheresis:

1. Targeted therapy, epigenetic therapy, or treatment with an investigational drug or used an invasive investigational medical device within 14 days or at least 5 half-lives, whichever is less.
2. Monoclonal antibody treatment for multiple myeloma within 21 days.
3. Cytotoxic therapy within 14 days.
4. Radiotherapy within 14 days.
5. Participated in other clinical trials within 30 days.

   8. Toxicity from previous anticancer therapy must resolve to baseline levels or to Grade 1 or less except for alopecia or peripheral neuropathy.

   9. With central nervous system involvement. 10. Serious underlying medical condition, such as:

a. Evidence of serious active viral, bacterial, or uncontrolled systemic fungal infection b. Active or unstable autoimmune diseases or autoimmune diseases that have been suffered within 3 years and have the possibility of recurrence c. Overt clinical evidence of dementia or altered mental status

11. Pregnant or breast-feeding, or planning to become pregnant while enrolled in this study or within 100 days after receiving study treatment.

12. Plans to father a child while enrolled in this study or within 100 days after receiving study treatment.

13. With obvious hemorrhagic tendency such as gastrointestinal hemorrhage, coagulation disorders and hypersplenism 14. Oxygen is needed to maintain sufficient blood oxygen saturation(≥95%) 15. Suffer from chronic diseases that require treatment with systemic corticosteroids or other immunosuppressive agents ,Received a cumulative dose of corticosteroids equivalent to ≥20 mg/day of prednisone within 7 days prior to apheresis 16. CNS diseases with clinical significance in the past or at the time of screening 17. Vaccinated with live, attenuated vaccine within 4 weeks prior to apheresis 18. Major surgery within 2 weeks prior to apheresis, or has surgery planned during the study or within 2 weeks after study treatment administration. (Note: subjects with planned surgical procedures to be conducted under local anesthesia may participate.) 19. Known life threatening allergies, hypersensitivity, or intolerance to LCAR-T2C CAR-T cells or its excipients, including DMSO (refer to Investigator's Brochure) 20. Presence of any condition that, in the opinion of the investigator, would prohibit the patient from undergoing treatment under this protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 30 days post infusion
  DLT assessed by NCI-CTCAE 5.0
Adverse events | 90 days post infusion
  Incidence and severity of adverse events as assessed by NCI-CTCAE 5.0
Recommended Phase II dose (RP2D) | 30 days post infusion
  RP2D established through ATD+BOIN design and the DLTs occurring following CAR T-cell infusion
Concentration of PK CAR positive T cells in peripheral blood and bone marrow | 2 years post infusion
  PK CAR positive T cells in peripheral blood, PK CAR transgene levels in peripheral blood, PK CAR positive T cells in bone marrow and PK CAR transgene levels in bone marrow.
Anti-drug antibody | 2 years post infusion
  Anti-drug antibody (ADA) will be conducted on blood sample for immune response analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Hu, MD/PhD, Principal Investigator — Beijing Boren Hospital
Locations (1):
- Beijing Boren Hospital, Beijing, Beijing Municipality, China